CLINICAL TRIAL: NCT00004887
Title: A Randomized Phase III Comparative Study of Paclitaxel With Carboplatin Versus Mitomycin, Ifosfamide, Cisplatin (MIC) Chemotherapy in Inoperable Advanced Stage Non-Small Cell Lung Cancer
Brief Title: Paclitaxel and Carboplatin Chemotherapy Compared With Standard Chemotherapy in Treating Patients With Stage III or Stage IV Non-small Cell Lung Cancer That Cannot Be Removed During Surgery
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Christie NHS Foundation Trust (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000067562; CHNT-PC/MIC; EU-99046
Record Dates: First submitted 2000-03-07; First posted 2003-07-24 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2000-03

CONDITIONS: Lung Cancer
Keywords: stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Cisplatin; Ifosfamide; Mitomycin; Paclitaxel; Vinblastine

INTERVENTIONS:
Drug: carboplatin
Drug: cisplatin
Drug: ifosfamide
Drug: mitomycin C
Drug: paclitaxel
Drug: vinblastine sulfate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known whether paclitaxel and carboplatin is more effective than standard chemotherapy for advanced non-small cell lung cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of paclitaxel and carboplatin chemotherapy with that of standard chemotherapy in treating patients who have stage III or stage IV non-small cell lung cancer that cannot be removed during surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the one and two year survival of patients with inoperable advanced non-small cell lung cancer treated with paclitaxel and cisplatin versus standard platinum therapy.
* Compare the toxic effects of these two regimens in this patient population.
* Compare the performance status, tumor response, and quality of life in these patients after these treatment regimens.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to center, stage of disease (IIIA vs IIIB vs IV), or performance status (ECOG O vs 1 vs 2 vs 3).

Patients are randomized to one of two treatment arms:

* Arm I: Patients receive paclitaxel IV over 3 hours, followed by carboplatin IV over 30 minutes on day 1.
* Arm II: Patients receive mitomycin IV, ifosfamide IV over 3 hours, and cisplatin IV over 1 hour on day 1 OR mitomycin IV, vinblastine IV, and cisplatin IV over 4 hours on day 1.

Treatment continues every 3 weeks for up to 4 courses in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed before each treatment course.

Patients are followed for survival.

PROJECTED ACCRUAL: Approximately 300 patients (150 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed inoperable advanced non-small cell lung cancer

  * Stage IIIA, IIIB, or IV
  * Not eligible for curative radiotherapy or surgery
* Measurable or evaluable disease

  * No bony lesions as only site of measurable disease
* No symptomatic brain metastases

PATIENT CHARACTERISTICS:

Age:

* Over 18

Performance status:

* ECOG 0-2 (ECOG 3 allowed in some cases)

Life expectancy:

* At least 12 weeks

Hematopoietic:

* WBC at least 3,000/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 2 times upper limit of normal (ULN)
* AST or ALT no greater than 3 times ULN (no greater than 5 times ULN for liver metastases)

Renal:

* Creatinine normal OR
* Creatinine clearance at least 60 mL/min

Other:

* Not pregnant
* Fertile patients must use effective contraception during and for 3 months after study
* No active infection
* No other serious systemic disorder that would preclude compliance
* No second malignancy except carcinoma in situ of the cervix or adequately treated basal cell skin cancer
* No peripheral neuropathy, significant neurological disorders (e.g., seizures), or psychiatric disorders

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics
* Prior radiotherapy allowed if measurable disease outside of irradiated field

Surgery:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-01

CONTACTS AND LOCATIONS:
Overall Officials: Nick Thatcher, PhD, FRCP, Study Chair — The Christie NHS Foundation Trust
Locations (1):
- Christie Hospital N.H.S. Trust, Manchester, England, United Kingdom